CLINICAL TRIAL: NCT03956784
Title: Impact of E-assisted Connected Follow up on the Delay of Management of Postoperative Complications in Digestive Surgery
Brief Title: E-assisted Follow up Diagnosis of Post Operative Digestive Complications
Acronym: SURGICONNECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 69HCL19_0343
Record Dates: First submitted 2019-05-15; First posted 2019-05-21 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Post-operative Complications After Colorectal Surgery; Post-operative Complications After Gastric Surgery; Post-operative Complications After Bariatric Surgery
Keywords: Bariatric surgery; Colorectal surgery; Gastric surgery; One day surgery; Post-operative complications; Follow-up care via Mobile App

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- E-assessed follow up (Experimental): Patients undergoing colorectal surgery (colectomy, sigmoidectomy, proctectomy, digestive stoma closure), bariatric or gastric, for whom an early discharge has been programmed, and followed by a connected application and a nursing logistics platform at home.
  Interventions: Device: E-assessed clinical and biological follow up
- Standard home follow-up care (Other): Patients undergoing surgery for colorectal surgery (colectomy, sigmoidectomy, proctectomy, digestive stoma closure), bariatric or gastric surgery, for whom an early discharge has been programmed, and followed by usual way.
  Interventions: Other: Usual at home follow up

INTERVENTIONS:
Device: E-assessed clinical and biological follow up — Clinical questionnaire: self-evaluation of pain (0 to 10), resumption of transit, bleeding, fever, pulse. In case of no filling, the patient is contacted.
  An automatic alert system is defined and divide the patient according to three situations:
  * Normal situation
  * Situation requiring the nurse to call back the patient and contact the surgeon if the assessment requires medical advice
  * Disturbing situation requiring contact of the first-line surgeon if a potentially serious event is suspected. Each speaker's place is described for each item in the detailed protocols
  Biological questionnaire:
  Biological monitoring (blood count, Ionogram, C-Reactive Protein, urea, creatinine) is performed on D1, D3 and D7.
  All information is accessible in real time by the surgeon who receives notifications by email and on his smartphone in case of clinical or biological abnormality on patient monitoring.
  Arms: E-assessed follow up
Other: Usual at home follow up — An information sheet on the clinical parameters to be monitored will be given to patients and will include the following information:
  1. Immediate complications and warning signs:
     * Tachycardia> 120 bpm
     * Dyspnea
     * Rectorragies and / or melena
     * Vomiting with or without presence of blood
     * Major abdominal pain (visual analogue scale> 6/10)
     * Fever> 38
  2. Management to deal with complications: call the service and / or the surgeon
  3. Actions to be performed by the patient after the exit:passage of the nurse during 10 days for anticoagulant morning and evening (identical in both study groups)
  Each patient will be given a prescription to perform a C-Reactive Protein assay on D1, D3 and D7, similarly.
  Arms: Standard home follow-up care

SUMMARY:
Postoperative management in digestive surgery has been modernized thanks to improved rehabilitation measures. These measures include an earlier refeeding, mobilization, restriction of infusions (out of a total of 22) and showed their benefit in colorectal, gastric and bariatric surgery. It is thus possible to perform sleeve gastrectomy, bypass, restorations of digestive continuity and colectomies with early discharge or one day surgery.

The most serious complications (fistula, sepsis) occur in the first 10 days postoperatively with an average readmission rate of 10%. Their screening is based on clinical signs (tachycardia, pain) or biological (C-Reactive Protein (CRP) assay on Day 3 or Day 4). It is important to manage these complications early so that their morbidity is lower, resulting in shorter stays and less severity.

The monitoring and safety of patients discharged early are therefore essential and for the moment poorly codified, ranging from simple nursing to follow-up via a health provider. Recently, coordination structures including nurse platform and smartphone follow up app have emerged. Thanks to this system, the patient collects his own history and biological results which allows him to be monitored continuously, as in the hospital. In case of no filling or sign of complication, the nurse platform contacts the patient.

This connected follow-up would make it possible to reinforce the safety of the patient discharged early after a complex digestive procedure performed on an outpatient basis. Its benefit has been poorly evaluated but it is however more and more used by surgeons convinced of its interest especially as it goes in the direction of the development of the outpatient activity requested by the High Authority of Health with economic benefits interesting also the administration of the care structures.

The purpose of the investigator's study is to evaluate the impact of e-assessed follow-up during 10 days after surgery compared to a conventional follow-up. The hypothesis is that this connected follow-up would allow earlier detection of complications requiring rehospitalization (within 48 hours), resulting in faster and less severe treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, age ≥18 years
* Patient hospitalized for colorectal, gastric or bariatric surgery
* Patient for whom an outpatient or enhanced recovery after surgery is performed (expected discharge no later than 4 days after surgery)
* Patient with a computer, tablet or mobile connected to internet
* Patient who agrees to be included in the study and who signs the informed consent form,
* Patient affiliated with a healthcare insurance plan.

Exclusion Criteria:

* Minor patient
* Patient who does not understand French, under supervision or guardianship
* Mentally unbalanced patients or unable to follow the instructions of a connected follow-up, from the point of view of the investigator
* Patient who is unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2020-06-23 (Actual); Primary Completion 2025-02-19 (Actual); Study Completion 2025-02-19 (Actual)

PRIMARY OUTCOMES:
Time required for the management of post-operative complications requiring rehospitalization | Within 6 months after surgery
  Number of hours between discharge from hospitalization after digestive surgery and readmission for hospitalization during which medical, surgical, radiological or endoscopic treatment is performed.

SECONDARY OUTCOMES:
Severe postoperative complication rate | Within 30 days after surgery
  Rate of medical and surgical (> or = grade 3) complications within 30 days after surgery using the Dindo-Clavien classification, described as:
  Grade I = Any deviation from the normal postoperative course. Grade 2 = Requiring pharmacological treatment with drugs other than such allowed for grade I complications.
  Grade III = Requiring surgical, endoscopic or radiological intervention, not under (Grade IIIa) or under general anesthesia (Grade IIIb) Grade IV = Life-threatening complication with single organ (Grade IVa) or Multiorgan dysfunction (Grade IVb) Grade V = Death of a patient.
Early overall complication rate | Within 30 days after surgery
  Rate of medical and surgical complications (each grade) within 30 days after surgery using the Dindo-Clavien classification
Type of early complications | Within 30 days after surgery
  Type (medical or surgical) of late complications (after 30 days) for each procedure according to the Dindo-Clavien classification
Severity of early complications | Within 30 days after surgery
  Severity of late complications (after 30 days) for each procedure according to the Dindo-Clavien classification
Late overall complication rate | Within 6 months after surgery
  Rate of medical and surgical complications (each grade) within 6 months after surgery using the Dindo-Clavien classification
Type of late complications | Within 6 months after surgery
  Type (medical or surgical) of late complications (after 6 months) for each procedure according to the Dindo-Clavien classification
Severity of late complications | Within 6 months after surgery
  Severity of late complications (after 6 months) for each procedure according to the Dindo-Clavien classification
Postoperative mortality | Within 30 days and 6 months after surgery
  Number of patients who died within 30 days and 6 months after surgery
Readmission of patient | Within 30 days and 6 months after surgery
  Number of patients readmitted within 30 days and 6 months after surgery.
Quality of life assessed with SF36 questionnaire | Before surgery and at 10 and 30 days after surgery
  Before surgery and at 10 and 30 days after surgery, according to the SF36 (Short Form (36) Health Survey) questionnaire.
  This questionnaire taps eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/tiredness, and general health perceptions. It also includes a single item that provides an indication of a perceived change in health.
Quality of life assessed with GIQLI questionnaire | Before surgery and at 10 and 30 days after surgery
  Before surgery and at 10 and 30 days after surgery, according to the GIQLI (Gastrointestinal Quality of Life index) questionnaire.
  This questionnaire consists of 36 items exploring 5 dimensions or subscales: symptoms, physical condition, emotions, social integration and the effect of any medical treatment. For each item, 5 responses will be proposed to the patients and for each answer, a score ranging from 0 to 4 (highest score = 144) will be assigned. A high score defines a more favorable health state.
Patient satisfaction: VAS | 10 days after surgery
  Satisfaction will be measured using a visual analog scale, rated from 0 (no satisfaction) to 10 (Perfect Satisfaction)
Patient sense of security | 10 days after surgery
  Sence of security will be measured using a visual analog scale, rated from 0 (no security felt) to 10 (Complete security felt Satisfaction)
Costs | 7 months post-inclusion
  Costs associated with the strategy including the Follow-up care via Mobile App compared to the standard follow-up care strategy.
Consequences | 7 months post-inclusion
  Consequences associated with the strategy including the Follow-up care via Mobile App compared to the standard follow-up care strategy.

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - Département de Chirurgie Digestive, Hôpital Michallon, CHU Grenoble, Grenoble
  - Service de Chirurgie Viscérale et Digestive, CH Emile Roux, Le Puy-en-Velay
  - Service de Chirurgie Générale, Digestive et de la Transplantation Hépatique, Hôpital de la Croix Rousse, Hospices Civils de Lyon, Lyon
  - Service de Chirurgie Digestive, Hôpital Edouard Herriot, Hospices Civils de Lyon, Lyon
  - Service de Chirurgie Digestive, Centre Hospitalier Lyon-Sud, Hospices Civils de Lyon, Pierre-Bénite
  - Service de Chirurgie Digestive et Oncologie Digestive, Hôpital Nord, CHU Saint-Etienne, Saint-Etienne